CLINICAL TRIAL: NCT00884390
Title: A Postauthorization Safety Surveillance Study Of Patients Switching To ReFacto AF From ReFacto Or Other Factor VIII Products In Usual Care Settings
Brief Title: Study Evaluating Safety Of Patients Switching To ReFacto AF In Usual Care Settings
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3082B2-4432
Record Dates: First submitted 2009-04-16; First posted 2009-04-20 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Hemophilia A
Keywords: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — recombinant factor VIII SQ; Factor VIII; Clinical Laboratory Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ReFacto AF (Experimental)
  Interventions: Drug: moroctocog alfa (AF-CC) (ReFacto AF); Procedure: Laboratory tests

INTERVENTIONS:
Drug: moroctocog alfa (AF-CC) (ReFacto AF) — Providing moroctocog alfa (AF-CC) as test article for use during this study.
Procedure: Laboratory tests — Laboratory samples are collected during study visits, in order to collect safety and efficacy data related to the administration of test article.

SUMMARY:
The study will be investigating safety in patients who switch to ReFacto AF from ReFacto and other Factor VIII products.

DETAILED DESCRIPTION:
The trial was terminated prematurely on 28 March 2013, due to the inability to recruit the planned number of subjects. The decision to terminate the trial was not based on any safety or efficacy concerns and agreement to close the study in March 2013 was agreed with EMA prior to closure activity.

ELIGIBILITY:
Inclusion Criteria:

* Male patients greater than or equal to 12 years of age with severe hemophilia A (FVIII:C less than 1%).
* Treatment history of greater than 150 EDs to prior recombinant or plasma-derived FVIII replacement products.
* Transitioning to ReFacto AF from ReFacto or other recombinant or plasma-derived FVIII replacement products.
* Serum albumin greater than or equal to the lower limit of normal (LLN).
* Platelet count greater than or equal to 100,000/µL.
* Prothrombin time (PT) less than or equal to1.25 × ULN, or international normalized ratio (INR) less than or equal to 1.5.
* HIV positive subjects must have a CD4 count greater than 200/µL and HIV viral load less than 200 particles/µL.

Exclusion Criteria:

* Presence of any bleeding disorder in addition to hemophilia A.
* A positive FVIII inhibitor, according to the local laboratory, at screening; or any Bethesda Inhibitor Titer greater than 0.6, regardless of the normal range for the testing laboratory.
* Treated with immunomodulatory therapy (including Immune Tolerance Induction [ITI]) during the screening period.
* Prior exposure to moroctocog alfa (AF-CC).
* Known hypersensitivity to hamster protein.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2009-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (72):
- Pfizer Investigational Site, Vienna, Austria
- Belgium (3):
  - Pfizer Investigational Site, Brussels, Belgium
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Leuven
- Pfizer Investigational Site, Copenhagen, Denmark
- Finland (2):
  - Pfizer Investigational Site, Helsinki
  - Pfizer Investigational Site, Kuopio
- France (11):
  - Pfizer Investigational Site, Chambray-lès-Tours
  - Pfizer Investigational Site, Clermont-Ferrand
  - Pfizer Investigational Site, Le Chesnay
  - Pfizer Investigational Site, Le Kremlin-Bicêtre
  - Pfizer Investigational Site, Limoges
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Montmorency
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Paris
- Germany (17):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bonn
  - Pfizer Investigational Site, Bremen
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Frankfurt am Main
  - Pfizer Investigational Site, Fulda
  - Pfizer Investigational Site, Halle
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Heidelberg
  - Pfizer Investigational Site, Homburg
  - Pfizer Investigational Site, Leipzig
  - Pfizer Investigational Site, Magdeburg
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Münster
  - Pfizer Investigational Site, Rostock
  - Pfizer Investigational Site, Stuttgart
  - Pfizer Investigational Site, Wiesbaden
- Pfizer Investigational Site, Athens, Greece
- Pfizer Investigational Site, Budapest, Hungary
- Italy (8):
  - Pfizer Investigational Site, Treviso, Castelfranco Veneto
  - Pfizer Investigational Site, Ivrea, Italy
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Pavia
  - Pfizer Investigational Site, Perugia
  - Pfizer Investigational Site, Udine
- Netherlands (3):
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Groningen
  - Pfizer Investigational Site, Utrecht
- Pfizer Investigational Site, Bucharest, Romania
- Spain (15):
  - Pfizer Investigational Site, A Coruña, A Coruna
  - Pfizer Investigational Site, Ávila, Avila
  - Pfizer Investigational Site, Palma de Mallorca, Balearic Islands
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Puerto Real, Cadiz
  - Pfizer Investigational Site, Málaga, Malaga
  - Pfizer Investigational Site, Madrid, Spain
  - Pfizer Investigational Site, Valencia, Valencia
  - Pfizer Investigational Site, Zaragoza, Zaragoza
  - Pfizer Investigational Site, Almería
  - Pfizer Investigational Site, Cadiz
  - Pfizer Investigational Site, Cáceres
  - Pfizer Investigational Site, Granada
  - Pfizer Investigational Site, Málaga
  - Pfizer Investigational Site, Valladolid
- Sweden (3):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Stockholm
- United Kingdom (5):
  - Pfizer Investigational Site, Birmingham, England
  - Pfizer Investigational Site, London, England
  - Pfizer Investigational Site, Edinburgh, Scotland
  - Pfizer Investigational Site, Bangor, Wales
  - Pfizer Investigational Site, Manchester

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3082B2-4432&StudyName=Study%20Evaluating%20Safety%20Of%20Patients%20Switching%20To%20ReFacto%20AF%20In%20Usual%20Care%20Settings

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two hundred and eight (208) participants were enrolled into the study (146 participants into the ReFacto Switch group [Cohort 1: participants who switched from ReFacto to ReFacto AF] and 62 participants into the Other Switch group [Cohort 2: participants who switched from other Factor VIII (FVIII) products other than ReFacto to ReFacto AF]).
Groups:
- ReFacto Switch: Participants who switched from ReFacto to ReFacto AF
- Other Switch: Participants who switched from other FVIII products other than ReFacto to ReFacto AF
Period: Overall Study
Arm/Group | ReFacto Switch | Other Switch
Started | 146 | 62
Completed | 123 | 54
Not Completed | 23 | 8
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Protocol Violation | 4 | 1
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Discontinuation of Study by Sponsor | 2 | 2
Not completed — Other | 11 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ReFacto Switch | Other Switch | Total
Number analyzed (Participants) | 146 | 62 | 208
Age, Customized [Number; unit: participants]
  12-17 years | 33 | 9 | 42
  18-65 years | 113 | 53 | 166
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 146 | 62 | 208

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Factor VIII Inhibitor Development
Description: Number of participants with clinically significant FVIII inhibitor development after switching from ReFacto to moroctocog alfa (AF-CC). Clinically significant inhibitors are defined as a central laboratory confirmed positive inhibitor (≥ 0.6 Bethesda unit (BU) using the Nijmegen modification of the Bethesda assay present at 2 consecutive blood draws within a 6-week interval) and within 28 days before the initial or within 28 days following the second positive FVIII inhibitor sample collection one of the following: the need for the participant to administer alternative hemostatic products in order to achieve sufficient efficacy, or ≥2 adverse event reports of decreased drug effect (or other adverse event indicating a decrease in the efficacy of the test article). The blood sample collection for these results must also be between the date of first dose of study medication and 28 days after the last dose of study medication.
Time Frame: 100 exposure days to study medication (approx. 2 years)
Population: All enrolled participants who took at least 1 dose of ReFacto AF study drug were included in the safety and efficacy analyses.
Measure: Number (95% Confidence Interval); unit: Number of participants
Arm/Group | ReFacto Switch | Other Switch
Number analyzed (Participants) | 146 | 62
Number of participants | 0 [0.00 to 2.49] | 0 [0.00 to 5.78]

2. Secondary Outcome: Annualized Bleeding Rates (ABRs)
Description: An ABR for each participant will be calculated as the number of bleeds requiring administration of FVIII replacement product (taken from the Infusion Log Diary case report form), divided by his total therapy duration (in days), then multiplied by 365.25.
Time Frame: 100 exposure days to study medication (approx. 2 years)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of bleeds
Groups:
- Annualized Bleed Rate: ABR by regimen at baseline is summarized for all participants for on-demand regimen, preventive regimen and prophylaxis regimen, respectively
Arm/Group | Annualized Bleed Rate
Number analyzed (Participants) | 208
Number of bleeds
  On-demand regimen (N=52) | 28.35 (18.781)
  Preventive regimen (N=2) | 1.08 (1.528)
  Primary or secondary prophylaxis regimen (N=154) | 8.43 (17.362)

3. Secondary Outcome: Response Assessment of First On-demand Treatment of New Bleeds
Description: A 4-point scale of assessment of 'on-demand' treatment (administration of an unscheduled bolus infusion of Refacto-AF to stop bleeding) is defined as:
  * Excellent: Definite pain relief and/or improvement in signs of bleeding starting within 8 hours after an infusion, with no additional infusion administered.
  * Good: Definite pain relief and/or improvement in signs of bleeding starting within 8 hours after an infusion, with at least one additional infusion administered for complete resolution of the bleeding episode; or, Definite pain relief and/or improvement in signs of bleeding starting after 8 hours following the infusion, with no additional infusion administered.
  * Moderate: Probable or slight improvement starting after 8 hours following the infusion, with at least one additional infusion administered for complete resolution of the bleeding episode.
  * No Response: No improvement at all between infusions or during the 24-hour interval following an infusion, or condition worsens.
Time Frame: 100 exposure days to study medication (approx. 2 years)
Population: as for outcome 1
Measure: Number; unit: Number of observations
Groups:
- First Infusion Per Bleed: Includes the first infusion for an associated bleeding episode
Arm/Group | First Infusion Per Bleed
Number analyzed (Participants) | 156
Number of observations
  Excellent | 1650
  Good | 1031
  Moderate | 191
  No response | 26
  Data Not Recorded | 343
  Total | 3241

4. Secondary Outcome: Number of ReFacto AF Infusions to Treat Each New Bleed
Description: The Infusion Log Diary case report form (CRF) was used to determine the number of test article infusions administered to treat a bleed. This was calculated by adding the initial (on-demand) infusion to any subsequent (on-demand) infusions for the same bleed (same bleed start date/time).
Time Frame: 100 exposure days to study medication (approx. 2 years)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Infusions
Groups:
- All Participants With Bleeds: Includes any infusion with an associated bleeding episode, regardless of the reason for treatment indicated on the case report form
Arm/Group | All Participants With Bleeds
Number analyzed (Participants) | 156
Number of Infusions
  Excellent | 1.1 (0.66)
  Good | 1.4 (1.45)
  Moderate | 2.0 (1.63)
  No response | 2.5 (2.60)
  Data Not Recorded | 1.3 (1.55)

5. Secondary Outcome: Number of Bleeding Episodes Occurring ≤48 Hours After a Prophylaxis Infusion
Description: First, the bleed start time from the Infusion Log Diary CRF was used to determine the number of breakthrough bleeds that occurred ≤48 hours after an infusion marked as "Prophylaxis" (which had no associated bleed). If there was more than 1 bleed location (ie, ankle and joint) with identical bleed start date and time, it was treated as 1 bleed occurrence. If a response was given, or if a bleed time was given, but "On Demand" was not listed as "treatment type", it was still counted as an on-demand bleed for analyses/summaries. Bleeding episodes were not categorized as spontaneous (atraumatic) or traumatic.
Time Frame: 100 exposure days to study medication (approx. 2 years)
Population: as for outcome 1
Measure: Number; unit: bleeds
Groups:
- Participants Who Received at Least One Prophylactic Infusion: Participants who had at least one prophylaxis dose, and at least one bleed.
Arm/Group | Participants Who Received at Least One Prophylactic Infusion
Number analyzed (Participants) | 108
bleeds | 96

6. Secondary Outcome: Number of Participants With Breakthrough Bleeds
Description: The number of participants with any breakthrough bleed was reported.
Time Frame: 100 exposure days to study medication (approx. 2 years)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Participants Who Received at Least One Prophylactic Infusion
Number analyzed (Participants) | 108
participants | 33

7. Secondary Outcome: Total Factor Consumption (TFC) Following a Non-prophylaxis Regimen at Baseline for All Participants
Description: The total amount (in International Units [IU]) infused for each test article infusion recorded in the Infusion Log Diary CRF was summed to calculate the TFC for each participant.
Time Frame: 100 exposure days to study medication (approx. 2 years)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: International Units (IU)
Groups:
- All Participants: All enrolled participants following a non-prophylaxis regimen at baseline.
Arm/Group | All Participants
Number analyzed (Participants) | 54
International Units (IU)
  On demand (n=50) | 115451.5 (67186.92)
  Preventive (n=43) | 35156.8 (40690.91)
  Prophylaxis (n=19) | 73001.9 (66969.64)
  Not specified (n=54) | 39268.3 (65013.77)
  Total (n=54) | 199848.9 (79308.82)

8. Secondary Outcome: TFC Following a Prophylaxis Regimen at Baseline for All Participants
Description: The total amount (in IU) infused for each test article infusion recorded in the Infusion Log Diary CRF was summed to calculate the TFC for each participant.
Time Frame: 100 exposure days to study medication (approx. 2 years)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | All Participants
Number analyzed (Participants) | 154
IU
  On Demand (n=98) | 26063.4 (32876.96)
  Preventive (n=65) | 22498.8 (29987.52)
  Prophylaxis (n=143) | 165124.6 (88373.55)
  Not specified (n=154) | 43812.8 (67588.23)
  Total (n=154) | 223224.8 (86493.58)

9. Secondary Outcome: Average Infusion Dose
Description: The average infusion dose for each participant was calculated as his total factor consumption (in IU) divided by the number of infusions administered. Summary statistics were reported for both of these variables separately for those participants classified at baseline as following an on-demand regimen, and for those on a primary or secondary prophylaxis regimen.
Time Frame: 100 exposure days to study medication (approx. 2 years)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU
Groups:
- Participants Following a Non-prophylaxis Regimen at Baseline: All enrolled participants following an on-demand or preventive regimen at baseline
- Participants Following a Prophylaxis Regimen at Baseline: All enrolled participants following a prophylaxis regimen at baseline
Arm/Group | Participants Following a Non-prophylaxis Regimen at Baseline | Participants Following a Prophylaxis Regimen at Baseline
Number analyzed (Participants) | 54 | 154
IU | 2326.8 (691.31) | 2290.3 (701.36)

10. Secondary Outcome: Incidence of Less-than-expected-therapeutic Effect (LETE) in the On-demand Setting
Description: The calculation of incidence of on-demand LETE used the number of bleeds identified as, or with a result of, LETE as the numerator (from the On Demand LETE CRF), and the denominator was the number of bleeding episodes treated in an on-demand setting. This denominator could include new bleeding episodes in prophylaxis participants breakthrough bleeds), and if subsequent on-demand doses for such a bleed met the on-demand LETE criteria, then an on-demand LETE was reported.
Time Frame: 100 exposure days to study medication (approx. 2 years)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of bleeds LETE
Groups:
- All Participants With at Least One Bleed: All enrolled participants with at least one bleed.
Arm/Group | All Participants With at Least One Bleed
Number analyzed (Participants) | 208
percentage of bleeds LETE | 0.06 [0.01 to 0.22]

11. Secondary Outcome: Incidence of Less-than-expected-therapeutic Effect (LETE) in the Prophylaxis Setting
Description: The calculation of incidence of prophylaxis LETE used the number of bleeds identified as, or with a result of, LETE as the numerator (from the Prophylactic LETE CRF), and the denominator was the number of routine prophylaxis infusions. Each infusion was classified in the infusion log ("Prophylaxis/ On Demand/ Preventive"), and participants were instructed to select "On Demand" if the infusion was to treat a bleed, even if the participant typically followed a prophylaxis regimen. Only the infusions classified as "Prophylaxis" were counted in this denominator.
Time Frame: 100 exposure days to study medication (approx. 2 years)
Measure: Number (95% Confidence Interval); unit: percentage of bleeding episodes
Groups:
- All Participants With at Least One Prophylaxis Infusion: All enrolled participants with at least one prophylaxis infusion
Arm/Group | All Participants With at Least One Prophylaxis Infusion
Number analyzed (Participants) | 208
percentage of bleeding episodes | 0.19 [0.12 to 0.28]

ADVERSE EVENTS:
Time Frame: Duration of participation in study
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- All Participants: The primary safety analysis was performed on all subjects who received at least 1 dose of ReFacto AF.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 20/208
Other Adverse Events (participants affected / at risk) | 90/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=208)
Factor VIII inhibition (Blood and lymphatic system disorders) | 5 (5)
Acute abdomen (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Intestinal haematoma (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1)
Acute tonsillitis (Infections and infestations) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1)
Septic arthritis streptococcal (Infections and infestations) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Anti factor VIII antibody positive (Investigations) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=208)
Nasopharyngitis (Infections and infestations) | 32 (44)
Influenza (Infections and infestations) | 13 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 (69)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 24 (86)
Limb injury (Injury, poisoning and procedural complications) | 15 (25)
Headache (Nervous system disorders) | 21 (47)

LIMITATIONS AND CAVEATS:
The study was terminated early by agreement with the EMA before full recruitment was attained, but this is not considered to affect the overall results and the ability of the study to address its objectives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.